CLINICAL TRIAL: NCT04025762
Title: An Open-label, Multi-centre, Randomised, Two-period, Crossover Study to Assess the Efficacy, Safety and Utility of 16 Week Day and Night Automated Closed-loop Glucose Control Under Free Living Conditions Compared to Sensor Augmented Insulin Pump Therapy in Older Adults With Type 1 Diabetes.
Brief Title: 24/7 Closed-loop in Older Subjects With Type 1 Diabetes
Acronym: DAN06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Chief Investigator, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN06
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia; Arrythmia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: An open-label, multi-centre randomised, two-period crossover study comparing day and night automated closed-loop glucose control with sensor-augmented pump therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day and night hybrid closed loop control (Experimental): The day and night hybrid closed-loop system (CamAPS FX) will consist of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
  Interventions: Device: Hybrid closed-loop system (CamAPS FX)
- Sensor augmented pump therapy (Active Comparator): The comparator will consist of Dana RS insulin pump (Sooil) and G6 real-time CGM sensor (Dexcom)
  Interventions: Device: Sensor augmented pump therapy

INTERVENTIONS:
Device: Hybrid closed-loop system (CamAPS FX) — Hybrid closed-loop system
  Arms: Day and night hybrid closed loop control
Device: Sensor augmented pump therapy — Sensor augmented pump therapy
  Arms: Sensor augmented pump therapy

SUMMARY:
The main objective of this open-label, multi-centre, randomised, crossover design study is to determine whether automated day and night closed-loop insulin delivery for 16 weeks under free living conditions is safer and more efficacious compared to sensor augmented insulin pump therapy in older adults with type 1 diabetes. The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L (70 and 180 mg/dl) as recorded by CGM. Secondary outcomes are the HbA1c, time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Measures of human factor assessments, cardiac arrhythmias and objective sleep quality assessment will also be evaluated in this study.

DETAILED DESCRIPTION:
No study thus far has specifically evaluated use of closed-loop insulin delivery in older adults with type 1 diabetes. During our previous closed-loop studies, if there is a communication failure between the algorithm device and the insulin pump, the pump is set to deliver pre-programmed basal insulin rates after about 30 to 60 minutes.The main objective of this study is to determine whether automated day and night closed-loop insulin delivery for 16 weeks under free living conditions is safer and more efficacious compared to sensor augmented insulin pump therapy in older adults with type 1 diabetes.

This is an open-label, multi-centre, randomised, crossover design study, involving a 4-6 week run-in period, followed by two 4 months study periods during which glucose levels will be controlled either by an automated closed-loop system or by sensor-augmented pump therapy in random order. A total of up to 42 adults (aiming for 36 completed subjects) aged 60 years and older with T1D on insulin pump therapy will be recruited through diabetes clinics and other established methods in participating centres. Subjects who drop out of the study within the first 6 weeks of the first intervention period will be replaced.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. Subjects will have regular contact with the study team during the home study phase including 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L (70 and 180mg/dl) as recorded by CGM. Secondary outcomes are the HbA1c, time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Measures of human factor assessments, cardiac arrhythmia and objective sleep quality assessment will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years and above
2. Type 1 diabetes as defined by WHO for at least 1 year or confirmed C-peptide negative
3. On insulin pump for at least 3 months with good knowledge of insulin self-adjustment
4. Treated with one of the U-100 rapid acting insulin analogues only (insulin Aspart, Lispro, Faster insulin Aspart but not Glulisine)
5. Willing to perform regular capillary blood glucose monitoring
6. HbA1c ≤ 10% (86 mmol/mmol) based on analysis from central laboratory or equivalent
7. Literate in English
8. Having a care partner who is aware of the subject's location and is trained to administer intramuscular glucagon and able to seek emergency assistance
9. Willing to wear closed-loop system at home and at work place
10. Willing to follow study specific instructions
11. Willing to upload pump and CGM data at regular intervals
12. Has access to WiFi

Exclusion Criteria:

1. Non-type 1 diabetes mellitus
2. Use of a closed-loop system within the last 30 days
3. Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
4. Use of any glucose-lowering agent (such as Pramlintide, Metformin, GLP-1 analogs) in the 3 months prior to enrolment or any use of SGLT2 inhibitors
5. Untreated coeliac disease, adrenal insufficiency or hypothyroidism
6. Known or suspected allergy against insulin
7. More than one episodes of severe hypoglycaemia as defined by American Diabetes Association in preceding 6 months
8. Random C-peptide > 200pmol/l with concomitant plasma glucose >4 mmol/l (72 mg/dl)
9. Lack of reliable telephone facility for contact
10. Total daily insulin dose >/= 2 IU/kg/day
11. Total daily insulin dose < 15 IU/day
12. Severe visual impairment
13. Severe hearing impairment
14. Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement
15. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which could potentially be used for localisation of the glucose sensor)
16. Subject is currently abusing illicit drugs
17. Subject is currently abusing prescription drugs
18. Subject is currently abusing alcohol
19. Subject has elective surgery planned that requires general anaesthesia during the course of the study
20. Subject is a shift worker with working hours between 10pm and 8am
21. Subject has a sickle cell disease, haemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
22. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
23. Subject diagnosed with current eating disorder such as anorexia or bulimia
24. Subject plans to use significant quantity of herbal preparations (use of over the counter herbal preparation for 30 consecutive days or longer period during the study) or significant quantity of vitamin supplements (four times the recommended daily allowance used for 30 consecutive days or longer period during the study) known to affect glucose metabolism and/or blood glucose levels during the course of their participation in the study
25. Subject not proficient in English (UK), or German (Austria)

Additional exclusion criteria specific for Austria

1. Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
2. Positive alcohol breath test.
3. Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 antibodies, anti-HIV2 antibodies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Schneider-Utaka AK, Hanes S, Boughton CK, Hartnell S, Thabit H, Mubita WM, Draxlbauer K, Poettler T, Hayes J, Wilinska ME, Mader JK, Narendran P, Leelarathna L, Evans ML, Hovorka R, Hood KK. Patient-reported outcomes for older adults on CamAPS FX closed loop system. Diabet Med. 2023 Sep;40(9):e15126. doi: 10.1111/dme.15126. Epub 2023 May 23. PMID 37171467
- [Derived] Boughton CK, Hartnell S, Thabit H, Mubita WM, Draxlbauer K, Poettler T, Wilinska ME, Hood KK, Mader JK, Narendran P, Leelarathna L, Evans ML, Hovorka R. Hybrid closed-loop glucose control compared with sensor augmented pump therapy in older adults with type 1 diabetes: an open-label multicentre, multinational, randomised, crossover study. Lancet Healthy Longev. 2022 Mar;3(3):e135-e142. doi: 10.1016/S2666-7568(22)00005-8. Epub 2022 Mar 7. PMID 35359882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew during the run-in period
Groups:
- Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy: The day and night hybrid closed-loop system (CamAPS FX) will consist of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
  Hybrid closed-loop system (CamAPS FX): Hybrid closed-loop system
- Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed-loop Control: The comparator will consist of Dana RS insulin pump (Sooil) and G6 real-time CGM sensor (Dexcom)
  Sensor augmented pump therapy: Sensor augmented pump therapy
Period: Run-in (3-4 Weeks)
Arm/Group | Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy | Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed-loop Control
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: Crossover Study Period 1 (16 Weeks)
Arm/Group | Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy | Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed-loop Control
Started | 20 | 17
Completed | 20 | 16
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: Washout Period (4 Weeks)
Arm/Group | Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy | Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed-loop Control
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0
Period: Crossover Study Period 2 (16 Weeks)
Arm/Group | Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy | Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed-loop Control
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy: Run-in period (3-4 weeks)
  16 weeks of day and night hybrid closed-loop system (CamAPS FX) consisting of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
  Hybrid closed-loop system (CamAPS FX): Hybrid closed-loop system
  Washout period (4 weeks)
- Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed Loop Control: Run-in period (3-4 weeks)
  16 weeks of the comparator consisting of Dana RS insulin pump (Sooil) and G6 real-time CGM sensor (Dexcom)
  Sensor augmented pump therapy: Sensor augmented pump therapy
  Washout period (4 weeks)
  16 weeks of day and night hybrid closed-loop system (CamAPS FX) consisting of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
  Hybrid closed-loop system (CamAPS FX): Hybrid closed-loop system
- Total: Total of all reporting groups
Arm/Group | Initial Use of Day and Night Hybrid Closed Loop Control Followed by Sensor Augmented Pump Therapy | Initial Use of Sensor Augmented Pump Therapy Followed by Day and Night Hybrid Closed Loop Control | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [63 to 70] | 67 [62 to 70] | 68 [63 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 16 | 15 | 31
  Austria | 4 | 2 | 6
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 38 [32 to 48] | 38 [32 to 48] | 38 [32 to 47]
Duration of pump therapy [Median (Inter-Quartile Range); unit: years] | 11 [8 to 16] | 9 [5 to 14] | 10 [7 to 15]
Charlson comorbidity index (lower value indicates less comorbidity burden) [Mean (Standard Deviation); unit: points on a scale (minimum 0 maximum 37)] | 4 (2) | 4 (1) | 4 (1)
Continuous glucose monitor user [Number; unit: participants] | 13 | 12 | 25
HbA1c, mmol/mol [Mean (Standard Deviation); unit: mmol/mol] | 58 (10) | 57 (9) | 57 (10)
HbA1c, % [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 7.5 (1.0) | 7.4 (0.9) | 7.4 (0.9)
Total daily insulin, units per day [Median (Inter-Quartile Range); unit: units/day] | 45.8 [38.3 to 51.1] | 40.0 [35.4 to 62.4] | 45.1 [36.8 to 57.2]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Time Spent in the Target Sensor Glucose Range During the 16 Week Intervention Period (%)
Description: Proportion of time spent in the target glucose range from 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on continuous glucose monitoring (CGM)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Mean (Standard Deviation); unit: % of time
Groups:
- Day and Night Hybrid Closed Loop Control: The day and night hybrid closed-loop system (CamAPS FX) will consist of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
  Hybrid closed-loop system (CamAPS FX): Hybrid closed-loop system
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 79.9 (7.9) | 71.4 (13.2)

2. Secondary Outcome: HbA1c at the End of the 16 Week Intervention Period (mmol/Mol)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
mmol/mol | 49.3 (7.9) | 52.1 (9.2)

3. Secondary Outcome: Proportion of Time Spent Below Target Glucose (3.9mmol/l) (70mg/dl) Based on CGM During the 16 Week Intervention Period (%)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 1.7 [1.3 to 2.4] | 1.7 [0.9 to 2.7]

4. Secondary Outcome: Proportion of Time Spent Above Target Glucose (10.0 mmol/l) (180 mg/dl) Based on CGM During the 16 Week Intervention Period (%)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 16.7 [11.4 to 23.9] | 21.4 [16.9 to 36.5]

5. Secondary Outcome: Average (mmol/L) of CGM Glucose Levels During the 16 Week Intervention Period
Time Frame: 16 weeks
Population: Crossover study design
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
mmol/L | 7.8 (0.7) | 8.5 (1.1)

6. Secondary Outcome: Proportion of Time With Glucose Levels < 3.5 mmol/l (63mg/dl) Based on CGM During the 16 Week Intervention Period (%)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 0.7 [0.5 to 1.1] | 0.7 [0.4 to 1.2]

7. Secondary Outcome: Proportion of Time With Glucose Levels in the Significant Hyperglycaemia (Glucose Levels > 16.7 mmol/l) (300mg/dl) Based on CGM During the 16 Week Intervention Period (%)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 0.5 [0.2 to 0.8] | 0.8 [0.2 to 2.8]

8. Secondary Outcome: Total Daily Insulin Dose During the 16 Week Intervention Period (Units/Day)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: units/day
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
units/day | 46.3 [36.9 to 53.5] | 42.9 [36.6 to 53.0]

9. Secondary Outcome: Standard Deviation (mmol/L) of CGM Glucose Levels During the 16 Week Intervention Period
Time Frame: 16 weeks
Population: Crossover study design
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
mmol/L | 2.6 (0.5) | 2.8 (0.6)

10. Other Pre Specified Outcome: The Proportion of Time of Use of the Closed-loop System at Home During the 16 Week Intervention Period (%)
Description: Utility evaluation
Time Frame: 16 weeks
Population: Closed-loop use was only measured during the closed-loop period.
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 0
% of time | 96.7 [95.1 to 98.0] |

11. Other Pre Specified Outcome: Cardiac Arrythmia Analysis
Description: Holter monitor data at the fourth month in the two treatment groups
Time Frame: 5-7 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Sleep Quality Assessment
Description: Sleep quality assessment using data collected by Actiwatch
Time Frame: 14 days
Reporting Status: Not Posted

13. Secondary Outcome: Proportion of Time With Glucose Levels < 3.0 mmol/l (54mg/dl) Based on CGM During the 16 Week Intervention Period (%)
Time Frame: 16 weeks
Population: Crossover study design
Measure: Median (Inter-Quartile Range); unit: % of time
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 36 | 37
% of time | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]

ADVERSE EVENTS:
Time Frame: Safety evaluation comprised the frequency of severe hypoglycaemia and diabetic ketoacidosis, and other adverse events or serious adverse events. Data were collected from recruitment until the final study visit, up to 10 months.
Description: Crossover study design
  Adverse events reported during the run-in period (pre-randomization) are reported for the whole study cohort and not by group as this was not determined at the time of the adverse event.
Groups:
- Day and Night Hybrid Closed Loop Control: 16 weeks of the day and night hybrid closed-loop system (CamAPS FX) which consists of:
  * Dana RS insulin pump (Sooil)
  * G6 real-time CGM sensor (Dexcom)
  * An unlocked android smartphone hosting the CamAPS FX app with Cambridge control algorithm
- Sensor Augmented Pump Therapy: 16 weeks of the comparator which consists of Dana RS insulin pump (Sooil) and G6 real-time CGM sensor (Dexcom)
- Run-in Period: 3-4 week run-in period with Dana RS insulin pump (Sooil) and G6 real-time CGM sensor (Dexcom)
- Washout Period: 4 week washout period between treatment periods when participants could continue to use the study devices with auto mode disabled or they could continue to use their pre-study devices
Arm/Group | Day and Night Hybrid Closed Loop Control | Sensor Augmented Pump Therapy | Run-in Period | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/37 | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/37 | 1/37 | 0/36
Other Adverse Events (participants affected / at risk) | 4/36 | 7/37 | 2/37 | 1/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day and Night Hybrid Closed Loop Control (N=36) | Sensor Augmented Pump Therapy (N=37) | Run-in Period (N=37) | Washout Period (N=36)
Death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unplanned hospital admission (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day and Night Hybrid Closed Loop Control (N=36) | Sensor Augmented Pump Therapy (N=37) | Run-in Period (N=37) | Washout Period (N=36)
Other (General disorders) | 4 (6) | 7 (9) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04025762/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04025762/SAP_001.pdf